CLINICAL TRIAL: NCT00144833
Title: A Phase III, Randomized, Controlled, Open-Label, Multicentre, Three Arm Study to Compare the Efficacy and Safety of a Dual-Boosted HIV-1 Protease Inhibitor Regimen of Fosamprenavir/Lopinavir/Ritonavir 1400mg/533mg/133mg Twice Daily and an Increased Dosage Regimen of FPV/RTV 1400mg/100mg BID Versus the Standard Dosage Regimen of FPV/RTV 700mg/100mg BID for 24 Weeks in Multiple-PI Experienced, HIV-Infected Adults Experiencing Virological Failure
Brief Title: Open Label Study of 908/RTV in Combination With Other PIs for the Treatment of Multi PI-Experienced HIV Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Incomplete data
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APV102002
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: HIV-1
Keywords: Protease inhibitors-experienced HIV-1 infected patients; Highly-resistant HIV-1; Dual boosted Pis; fosamprenavir; lopinavir
MeSH Terms: interventions — fosamprenavir; Ritonavir; BID protein, human; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fosamprenavir/ritonavir (700mg/100mg BID)
Drug: fosamprenavir/ritonavir (1400mg/100mg BID)
Drug: fosamprenavir/lopinavir/ritonavir (1400mg/533mg/100mg BID)

SUMMARY:
For HIV-infected individuals with highly resistant viruses, higher drug levels may be required to block the virus. This study investigates that concept by comparing the efficacy of standard fosamprenavir/ritonavir to an increased dose of boosted fosamprenavir and to a combination of fosamprenavir (increased dose)/lopinavir/ritonavir.

ELIGIBILITY:
Inclusion criteria:

* Multiple protease-inhibitors experienced HIV-1 infected individuals experiencing virological failure and who's virus is not fully resistant to boosted fosamprenavir and boosted lopinavir based on genotypic resistance tests.

Exclusion criteria:

* No full resistance to FPV/r or LPV/r
* Planned use of NNRTIs as part of the study salvage regimen
* Application of additional exclusion criteria as determined by physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-03

PRIMARY OUTCOMES:
The average area under the curve minus baseline [AAUCMB] in plasma HIV-1 RNA at 24 Weeks when each are administered in combination with an optimised background therapy, in a multiple PI-experienced population experiencing virological failure. | 24 weeks

SECONDARY OUTCOMES:
Efficacy (AAUCMB) at 48 weeks, safety, tolerability(incidence and nature of AEs and laboratory abnormalities) at week 24 and 48, CD4 change from baseline at week 24 and 48, and the steady-state plasma APV and LPV through concentrations. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (32):
- Australia (2):
  - GSK Clinical Trials Call Center, Darlinghurst, New South Wales
  - GSK Clinical Trials Call Center, Carlton, Victoria
- GSK Clinical Trials Call Center, Brussels, Belgium
- Canada (6):
  - GSK Clinical Trials Call Center, Vancouver, British Columbia
  - GSK Clinical Trials Call Center, Hamilton, Ontario
  - GSK Clinical Trials Call Center, Ottawa, Ontario
  - GSK Clinical Trials Call Center, Toronto, Ontario
  - GSK Clinical Trials Call Center, Montreal, Quebec
  - GSK Clinical Trials Call Center, Saint-Foy, Quebec
- France (7):
  - GSK Clinical Trials Call Center, Lagny-sur-Marne
  - GSK Clinical Trials Call Center, Paris
  - GSK Clinical Trials Call Centre, Paris
  - GSK Clinical Trials Call Center, Saint-Denis
  - GSK Clinical Trials Call Center, Strasbourg
  - GSK Clinical Trials Call Center, Toulon
  - GSK Clinical Trials Call Center, Vanouvre Les Nancy
- GSK Clinical Trials Call Center, Hamburg, Germany
- Greece (2):
  - GSK Clinical Trials Call Center, Athens
  - GSK Clinical Trials Call Center, Piraeus
- Italy (7):
  - GSK Clinical Trials Call Center, Liguria
  - GSK Clinical Trials Call Center, Lombardia
  - GSK Clinical Trials Call Center, Romagna
  - GSK Clinical Trials Call Center, Rome
  - GSK Clinical Trials Call Centre, Torino
  - GSK Clinical Trials Call Center, Toscana
  - GSK Clinical Trials Call Center, Veneto
- Spain (3):
  - GSK Clinical Trials Call Center, Barcelona
  - GSK Clinical Trials Call Center, Jerez de la Frontera
  - GSK Clinical Trials Call Center, Madrid
- United Kingdom (3):
  - GSK Clinical Trials call Center, Birmingham
  - GSK Clinical Trials Call Center, Brighton
  - GSK Clinical Trials Call Center, London